CLINICAL TRIAL: NCT01966822
Title: MULTICENTRE STUDY TO ASSESS CHANGES IN BONE MINERAL DENSITY OF THE SWITCH FROM PROTEASE INHIBITORS TO DOLUTEGRAVIR IN HIV-1-INFECTED SUBJECTS WITH LOW BONE MINERAL DENSITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSTEODOLU
Record Dates: First submitted 2013-10-07; First posted 2013-10-22 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: HIV-1 Infection
Keywords: Osteoporosis; Bone mineral density; Dual-energy X-ray absorptiometry; HIV infection; Dolutegravir; Integrase inhibitor
MeSH Terms: conditions — Osteoporosis; HIV Infections | interventions — dolutegravir; Protease Inhibitors; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dolutegravir 50mg (Experimental): Dolutegravir 50mg every 24 hours + Kivexa (ABC+3TC)
  Interventions: Drug: Dolutegravir, 50mg every 24 hours
- Protease Inhibitor/ritonavir (Active Comparator): Protease Inhibitor/ritonavir + Kivexa (ABC+3TC)
  Interventions: Drug: Protease Inhibitor/ritonavir

INTERVENTIONS:
Drug: Dolutegravir, 50mg every 24 hours — Dolutegravir, 50mg every 24 hours
  Arms: Dolutegravir 50mg
Drug: Protease Inhibitor/ritonavir — Protease Inhibitor/ritonavir
  Arms: Protease Inhibitor/ritonavir

SUMMARY:
Protease inhibitors (PI) have been associated with an acceleration of bone mineral density loss in HIV-infected individuals because of an enhanced osteoclast activity, although some controversial data have been also published. A first study suggest an increase of bone mineral density after switching from PI to raltegravir, the first generation integrase inhibitor, but there are no more data about this subject.

Based on data that PI decrease bone mineral density by accelerating osteoclast cells and that the discontinuation of this drugs could improve bone mineralization, we propose a randomized prospective multicenter study to assess the impact of switching from PI to dolutegravir on bone mineral density in patients with low bone mineral density receiving a PI-containing regimen. At the same time, the study will help to assess the antiviral efficacy and safety of a PI-sparing regimen including dolutegravir as a simplification strategy in virologically suppressed patients.

DETAILED DESCRIPTION:
The second generation integrase inhibitor dolutegravir has demonstrated good virological and immunological outcomes in antiretroviral-naive subjects, compared with efavirenz, (SPRING 1 study). As well, it is active against HIV strains resistant to first-generation inhibitors raltegravir and elvitegravir in heavily treatment-experienced patients (VIKING study).

Additionally, it was safe and well tolerated after two years of use. It is administered once daily with no need for boosting, no food requirements and has a long half-life. The easy posology and its pharmacokinetics, together with the antiviral potency, make this drug a good alternative as a simplification approach. However, no clinical data are available supporting the switch of protease inhibitors or no nucleoside reverse transcriptase inhibitors to dolutegravir in virologically suppressed HIV-treated subjects.

Protease inhibitors (PI) have been associated with an acceleration of bone mineral density loss in HIV-infected individuals because of an enhanced osteoclast activity, although some controversial data have been also published. A first study suggest an increase of bone mineral density after switching from PI to raltegravir, the first generation integrase inhibitor, but there are no more data about this subject.

Based on data that PI decrease bone mineral density by accelerating osteoclast cells and that the discontinuation of this drugs could improve bone mineralization, we propose a randomized prospective multicenter study to assess the impact of switching from PI to dolutegravir on bone mineral density in patients with low bone mineral density receiving a PI-containing regimen. At the same time, the study will help to assess the antiviral efficacy and safety of a PI-sparing regimen including dolutegravir as a simplification strategy in virologically suppressed patients.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected patients over 18 years.
2. In current antiretroviral therapy with abacavir and lamivudine (Kivexa) plus ritonavir-boosted PI, at least 6 months.
3. Viral suppression (HIV RNA <50 copies / ml) for at least 12 months.
4. T-score ≤ -1 evaluated by DEXA (done in the last 6 months).
5. Signed informed consent.
6. In potential childbearing women, commitment to use barrier contraceptive method throughout the study.

Exclusion Criteria:

1. Suspected or documented resistance to integrase inhibitors or reverse transcriptase inhibitors, nucleoside analogues.
2. Osteoporosis / osteopenia secondary (testosterone deficiency, thyroid disease ...), except vitamin D deficiency
3. Treatment with bisphosphonates in the last 6 months.
4. Have used integrase inhibitors
5. Pregnant or breastfeeding.
6. Patients with alanine aminotransferase (ALT)> 5 times the upper limit of normal (ULN) or ALT ≥ 3 times ULN and bilirubin ≥ 1.5 times ULN (direct bilirubin> 35%)
7. Patients with severe hepatic dysfunction (Class B or C) according to the Child-Pugh classification
8. Patients infected with hepatitis B virus (HBV) who can not use entecavir or telbivudine.
9. Patients infected with hepatitis C virus (HCV) in which is expected to begin treatment during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Compare changes in Bone Mineral Density (BMO) measured by Dual-energy X-ray absorptiometry | From Baseline to week 48
Compare changes in femur T-score measured by DEXA | From Baseline to week 48
Compare changes in lumbar spine (L1-L4) T-score measured by DEXA | From Baseline to week 48

SECONDARY OUTCOMES:
HIV-1 viral load | Baseline
HIV-1 viral load | week 4
HIV-1 viral load | week 12
HIV-1 viral load | week 24
HIV-1 viral load | week 48
CD4+/CD8+ T lymphocytes count. | Baseline
CD4+/CD8+ T lymphocytes count. | week 4
CD4+/CD8+ T lymphocytes count. | week 12
CD4+/CD8+ T lymphocytes count. | week 24
CD4+/CD8+ T lymphocytes count. | week 48
Genotypic test if virological failure occurs. | From baseline to week 48
Compare changes in total cholesterol | at week 48 relative to baseline values
Compare changes in HDL cholesterol | at week 48 relative to baseline values
Compare changes in LDL cholesterol | at week 48 relative to baseline values
Compare changes in triglyceride levels. | at week 48 relative to baseline values
Compare changes in filtrate glomerular rate by MDRD equation | at week 48 relative to baseline values
Compare changes in creatinine | at week 48 relative to baseline values
Compare changes in albumine/creatinine ratio | at week 48 relative to baseline values
Compare changes in proteinuria/creatinine ratio | at week 48 relative to baseline values
Adverse events related to antiretroviral treatment (Toxicity). | From Baseline to week 48
Patient withdrawal | From Baseline to week 48
Compare changes in osteocalcin | at week 48 relative to baseline values
Compare changes in alkaline phosphatase | at week 48 relative to baseline values
Compare changes in telopeptide | at week 48 relative to baseline values

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - GermansTrias i Pujol Hospital, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid, Madrid